CLINICAL TRIAL: NCT02547259
Title: Influence of Negative or Painful Emotions in a Directed Forgetting Paradigm in Healthy Subjects and Patients With Schizophrenia
Brief Title: Influence of Emotion in a Test Run Forgetfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1108067; 2011-A00582-39 (Other: AFSSAPS)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia; Healthy Volunteer
Keywords: schizophrenia; memory; pain
MeSH Terms: conditions — Schizophrenia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- schizophrenic pain words test (Experimental): schizophrenic will have memory test with pain words on computer
  Interventions: Procedure: pain words test
- schizophrenic negative words test (Experimental): schizophrenic will have memory test with negative words on computer
  Interventions: Procedure: negative words test
- Healthy volunteer pain words test (Other): Healthy volunteer will have memory test with pain words on computer
  Interventions: Procedure: pain words test
- Healthy volunteer negative words test (Other): Healthy volunteer will have memory test with negative words on computer
  Interventions: Procedure: negative words test

INTERVENTIONS:
Procedure: pain words test — words to painful sense will be shown on a screen, one at a time for 5 seconds. Patient or healthy volunteer will need to retain them. Then these same words, mixed with others that patient/healthy volunteer will not learn, will again be displayed on the computer screen one at a time for 5 seconds. Upon the occurrence of a word, patient/healthy volunteer must press the 'L' key if they think they have learned the word or the "D" key on the keyboard if they feel that they have not learned this word.
  Arms: Healthy volunteer pain words test; schizophrenic pain words test
Procedure: negative words test — words to negative sense will be shown on a screen, one at a time for 5 seconds. Patient or healthy volunteer need to retain them. Then these same words, mixed with others that patient/healthy volunteer will not learn, will again be displayed on the computer screen one at a time for 5 seconds. Upon the occurrence of a word, patient/healthy volunteer must press the 'L' key if they think they have learned the word or the "D" key on the keyboard if they feel that they have not learned this word.
  Arms: Healthy volunteer negative words test; schizophrenic negative words test

SUMMARY:
Currently there is uncertainty on how schizophrenic patients feel pain. Pain has several components including cognitive behavior which allow humans to perceive it as a negative emotion. It is difficult to say precisely what are the differences in cognitive processing between the emotional component of pain and painless another negative emotion (eg fear). However, pain and negative emotion have some neural networks together and there are many common ways between emotional processing (pain or negative) and storing information (limbic system).

DETAILED DESCRIPTION:
The study is to go 1 time in hospital for memory test. These tests consist in:

* Group 1: words to painful sense will be shown on a screen, one at a time for 5 seconds. Patient or healthy volunteer will need to retain them. Then these same words, mixed with others that patient/healthy volunteer will not learn, will again be displayed on the computer screen one at a time for 5 seconds. Upon the occurrence of a word, patient/healthy volunteer must press the 'L' key if they think they have learned the word or the "D" key on the keyboard if they feel that they have not learned this word.
* Group 2: words to negative sense will be shown on a screen, one at a time for 5 seconds. Patient or healthy volunteer need to retain them. Then these same words, mixed with others that patient/healthy volunteer will not learn, will again be displayed on the computer screen one at a time for 5 seconds. Upon the occurrence of a word, patient/healthy volunteer must press the 'L' key if they think they have learned the word or the "D" key on the keyboard if they feel that they have not learned this word.

  15 schizophrenic will be included in group 1 and 15 other schizophrenics in group 2.

  15 Healthy volunteer will be included in group 1 and 15 other Healthy volunteer in group 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients:
* schizophrenic age 18 years to 55 years
* Stabilized, clinical and therapeutic point of view, since at least one month.
* Good knowledge of French
* Healthy volunteer
* age 18 years to 55 years
* Good knowledge of French
* Matching on age (± 5 years) and level of study patients

Exclusion Criteria:

* Patients
* History of head trauma, neurological disease with cerebral repercussion or not stabilized or serious physical illness causing pain> 3 months.
* Recent Amendment of psychotropic therapy (<1 month)
* Consumption of benzodiazepines long-term (negative effect on memory capacity)
* Troubles Related to the use of a psychoactive substance, as defined by the DSM IV (recent use, abuse, dependence or withdrawal).
* Healthy volunteer
* Consumption of benzodiazepines long-term (negative effect on memory capacity)
* Troubles Related to the use of a psychoactive substance, as defined by the DSM IV (recent use, abuse, dependence or withdrawal).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Retained words | Day 1
  Number of selected words and average time taken to recognize between healthy volunteers and schizophrenics (composite measure)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MASSOUBRE, MD-PhD, Principal Investigator — CHU SAINT-ETIENNE